CLINICAL TRIAL: NCT04170049
Title: The Effects of Sensory Stimulative Activities on Sleep Performance in Community-dwelling Older Adults : A Single-case Design
Brief Title: The Effects of Sensory Stimulative Activities on Sleep Performance in Elderly Adults: A Single-case Design
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 201903021RINA
Record Dates: First submitted 2019-11-18; First posted 2019-11-20 (Actual); Last update posted 2019-11-26 (Actual); Status verified 2019-04

CONDITIONS: Sleep Disturbance
MeSH Terms: conditions — Parasomnias

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Behavioral: The sensory stimulative activity interventions (Experimental)
  Interventions: Behavioral: Sensory Stimulative Activitiy ( proprioceptive intervention, music intervention )

INTERVENTIONS:
Behavioral: Sensory Stimulative Activitiy ( proprioceptive intervention, music intervention ) — Music intervention: Listening to soft music was found to be an effective method of relaxation, as indicated by a shift of the autonomic balance toward parasympathetic activity. Participants listen to preferred soft music for 30 minutes before sleeping. Proprioceptive intervention: The proprioceptive intervention can activate the parasympathetic nervous system through pathways of the central nervous system, providing calming effects that significantly reduce anxiety, hyperactivity and agitation in various populations.Participants do 10-minute joint compression exercise three times per day by themselves.

SUMMARY:
Older adults have a high prevalence of sleep disturbances, which negatively and severely impact their health and quality of life. Research indicated that 43% elderly outpatients in Taiwan have used benzodiazepine, which collectively led to great medical expenditure. Non-pharmacological treatments are highly recommended as first priority for sleep disturbance in practice. Music interventions have been reported to modulate the sympathetic nervous system and to improve the elderly's sleeping performance. Proprioceptive interventions can also activate the parasympathetic nervous system, providing calming effects and significantly reducing anxiety, hyperactivity and agitation in various populations. However, the effects of these intervention on the sleep disturbances in the elderly remain unclear. The research purpose is to investigate the effects of two sensory activities that are easily executed in everyday life - auditory (e.g. listening to the music before sleeping) and proprioceptive (e.g. joint compression exercises) interventions on improving the sleep performance of the elderly. Subjective sleeping quality assessment (Pittsburgh Sleep Quality Index & Insomnia Severity Index) and objective physiological records measured by actigraphy are used as outcome measures.

DETAILED DESCRIPTION:
In this single-case designs study, we will recruit six volunteering elderly with primary insomnia and use A-B-A-C-A-D design for 9 weeks including the three periods of baseline phases for 1 week(A), the music intervention phase for 2 weeks(B), the proprioceptive intervention phase for 2 weeks(C) and the combination phase for 2 weeks(D). The main outcome measures include the objective sleeping quality measured everyday by the actigraphy recording the sleeping performance and physiological data during sleep, and the subjective sleeping quality measured every week via the Pittsburgh Sleep Quality Index and the Insomnia Severity. The secondary outcome measures, including the Center for Epidemiologic Studies Depression Scale, Geriatric Anxiety Scale - Chinese Version and WHOQOL-BREF, will be assessed weekly. The above results will present in visually analyzing graphed data to compare the performance among different phases and to evaluate the impacts of different interventions. This study will aim to preliminary investigate the feasibility and effectiveness of the music intervention, the proprioception intervention and the combination of both approaches on improving the objective sleeping performance and the subjective sleeping quality of the elderly.

ELIGIBILITY:
Inclusion Criteria:

1. have experienced insomnia (PSQI>5 at screening;) for at least one month.
2. Over 65 years of age or older.

Exclusion Criteria:

1. psychiatric or neurological problems
2. a history of alcohol / drug abuse
3. Hearing impaired.

Min Age: 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Older Adult
Enrollment: 6 (Estimated)
Dates: Start 2019-04-01 (Actual); Primary Completion 2020-05-06 (Estimated); Study Completion 2022-04-01 (Estimated)

PRIMARY OUTCOMES:
ActiGraph GT9X | erveryday during 9 weeks
  The objective sleep quality (sleep quality, sleep total time, sleep latency, awakening time during sleep)
The Pittsburgh Sleep Quality Index | once a week during 9 weeks
  The Pittsburgh Sleep Quality Index (PSQI) is a self-report questionnaire that assesses sleep quality over a 1-month time interval. The measure consists of 19 individual items, creating 7 components that produce one global score, and takes 5-10 minutes to complete. Scoring of the answers is based on a 0 to 3 scale, whereby 3 reflects the negative extreme on the Likert Scale.
  A global sum of "5"or greater indicates a "poor" sleeper.
The Insomnia Severity Index | once a week during 9 weeks
  a brief instrument(7 items) that was designed to assess the severity of both nighttime and daytime components of insomnia.(Total score categories: 0-7 = No clinically significant insomnia, 8-14 = Subthreshold insomnia, 15-21 = Clinical insomnia (moderate severity), 22-28 = Clinical insomnia (severe)) It is available in several languages and is increasingly used as a metric of treatment response in clinical research.

SECONDARY OUTCOMES:
The Center for Epidemiologic Studies Depression Scale | once a week during 9 weeks
  The CES-D scale is a brief self-report scale designed to measure self-reported symptoms associated with depression experienced in the past week. The items of the scale are symptoms associated with depression which have been used in previously validated longer scales.Possible range of scores is zero to 60, with the higher scores indicating the presence of more symptomatology.
Geriatric Anxiety Scale - Chinese Version | once a week during 9 weeks
  The Geriatric Anxiety Scale is a 30-item self-report measure used to assess anxiety symptoms among older adults.Individuals are asked to indicate how often they have experienced each symptom during the last week, answering on a 4-point Likert scale ranging from "Not at all" (0) to "All the time" (3).
WHO Quality of Life-BREF (WHOQOL-BREF) | once a week during 9 weeks
  The WHOQOL-BREF instrument comprises 26 items, which measure the following broad domains: physical health, psychological health, social relationships, and environment. The WHOQOL-BREF is a shorter version of the original instrument that may be more convenient for use in large research studies or clinical trials.

CONTACTS AND LOCATIONS:
Locations (1):
- National Taiwan University, Taipei, Taiwan

IPD SHARING:
Plan to Share IPD: No